CLINICAL TRIAL: NCT01935726
Title: Pulmonary Fibrosis Contact Registry
Status: Completed | Type: Observational
Sponsor: National Jewish Health (Other)
Collaborators: Pulmonary Fibrosis Foundation (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Jeff Swigris, Associate Professor of Medicine, National Jewish Health
Other Study IDs: PCORI 4134
Record Dates: First submitted 2013-08-31; First posted 2013-09-05 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Pulmonary Fibrosis of Any Cause; Primary Supporters/Caretakers of Patients With Pulmonary Fibrosis
Keywords: Pulmonary fibrosis; Interstitial lung disease; Connective tissue disease; Chronic hypersensitivity pneumonitis; Idiopathic pulmonary fibrosis
MeSH Terms: conditions — Pulmonary Fibrosis; Lung Diseases, Interstitial; Connective Tissue Diseases; Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Pulmonary fibrosis patients or their caretaker/supporter: Patients with pulmonary fibrosis of any cause (idiopathic, related to connective tissue disease [e.g., rheumatoid arthritis, systemic sclerosis/scleroderma, dermato-/polymyositis, sjogren's syndrome], familial or genetic) or the primary supporter/caregiver of a patient with pulmonary fibrosis

SUMMARY:
As the name states, contact registries securely store contact information from groups of reasonably well-characterized patients (or primary supporters/caregivers) who are interested in being informed about ongoing or future research opportunities. Pulmonary fibrosis (PF) is a condition for which effective therapies have remained elusive, making drug trials and interventional research studies a mainstay in the PF arena over the last decade and for the foreseeable future. A PF Contact Registry will be a conduit to collect, analyze, and disseminate de-identified, group-level data on the clinical phenotypes of PF patients and will house contact information from patients who wish to be informed about research opportunities for which they may qualify. Data contained in the Registry will help inform research hypotheses and guide investigators as they develop research protocols by providing them with numbers of potential subjects who meet particular inclusion/exclusion criteria.

DETAILED DESCRIPTION:
Detailed information can be found at our website at www.pulmonaryfirbrosisresearch.org.

Who will be in the Registry?

Anyone who is at least 18 years of age, can read and understand English, and either

1. diagnosed with PF or
2. a primary supporter or caregiver of someone living with PF

How the Registry works

Patients with PF consent to be enrolled in the Registry and may consent to be contacted by Registry personnel about opportunities for them to participate in research studies. Some of these studies (e.g., "Observing the Effects of Supplemental Oxygen on Patients with Pulmonary Fibrosis") will be conducted by Dr. Swigris and his research team-these studies will be considered Registry-affiliated. Registry participants are free to enroll in any study they wish-whether Registry-affiliated or conducted by investigators not affiliated with the Registry-i.e., non-Registry-affiliated studies. It is assumed the investigators conducting those studies will adhere to regulations governing the protection of human subjects in research. Consider a hypothetical example: an investigator in Michigan is conducting a study of the effects of oral honey on PF-related cough and would like Registry participants to consider enrollment. The investigator would petition the Registry and, if approved by the Registry Oversight Committee, Registry personnel would contact potentially eligible Registry participants to inform them of the study. The participants would then decide whether or not to contact the investigator in Michigan to be considered for enrollment. The investigatory in Michigan would be responsible for discussing the study with any potential subject, obtaining informed consent and conducting the study. All of these fall outside the purview of the Registry or its personnel.

How subjects will enroll in the Registry

Eligible participants must fill out an intake questionnaire/consent form. Contact information provided to receive a questionnaire is not stored by the Registry Data Coordinating Center (DCC) or by the study coordinator. Subjects may obtain the intake questionnaire, complete it, and submit it four different ways:

* Complete the questionnaire/consent form and submit it online at https://dccweb.njhealth.org/sec/P3F_Swigris/Index.htm. Participants will be encouraged to print a copy for their records.
* Enter a mailing address onto an online form at http://pulmonaryfibrosisresearch.org/contact and have a hard copy mailed to the subject. Once a signed questionnaire/consent has been sent back to the study coordinator, a copy will be made and mailed back to the participant for his/her records.
* Fill out the form electronically at https://dccweb.njhealth.org/sec/P3F_Swigris/Index.htm and print a copy of the form, or print the form and fill it out by hand and mail or fax the completed questionnaire to the study coordinator who will then hand it off to the DCC at National Jewish Health. Participants will be encouraged to print a copy for their records.
* Call the study coordinator toll-free at 1-855-609-0010 and have him/her mail a hard copy of the questionnaire/consent form to the subject. Once a signed questionnaire/consent has been sent back to the study coordinator, a copy will be made and mailed back to the participant for his/her records.

ELIGIBILITY:
Inclusion Criteria:

* Anyone who self-reports a diagnosis of pulmonary fibrosis and is over 18 years of age will be included in the Registry.
* Anyone who self-reports being a primary supporter or caregiver of someone living with pulmonary fibrosis and is over the age of 18 will be included in the Registry.
* Whoever consents to be enrolled in the Registry will presumably be able to read and write in English.

Exclusion Criteria:

* Failure to meet inclusion criteria

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with pulmonary fibrosis of any cause (idiopathic, related to connective tissue disease [e.g., rheumatoid arthritis, systemic sclerosis/scleroderma, dermato-/polymyositis, sjogren's syndrome], familial or genetic) or the primary supporter/caregiver of a patient with pulmonary fibrosis
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2013-08; Primary Completion 2019-03-10 (Actual); Study Completion 2019-03-10 (Actual)

PRIMARY OUTCOMES:
Number enrolled | 20 years
  This is a contact registry. We will enroll as many patients and primary supporters/caretakers as possible.

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Swigris, DO, MS, Principal Investigator — National Jewish Health
Locations (1):
- National Jewish Health Interstitial Lung Disease Program, Denver, Colorado, United States